CLINICAL TRIAL: NCT06713330
Title: A 36-Month Prospective Randomized Clinical Pilot Trial Comparing Stainless Steel Crowns with Prefabricated Resin Crowns in Primary Molar Teeth
Brief Title: Comparing Stainless Steel Crowns with Prefabricated Resin Crowns in Primary Molar Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Patrick Ruck, Primary investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0022
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries
Keywords: Pediatric dentistry
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: The purpose of this 36-month prospective, randomized controlled, split-mouth pilot study, is to compare a new prefabricated resin crown material against the gold standard stainless steel crown in primary molars that require full coverage restorations. The results of this study can help determine if resin polymer crowns clinically perform like stainless steel crowns, and if they are an acceptable esthetic alternative treatment option for a full coverage restoration of a primary molar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SSC (Other): Experimental: 3M Stainless Steel Crowns. In this split-mouth design, subjects were randomly assigned to receive SSC in the left or right side of the mouth.
  Interventions: Device: 3M Stainless Steel Crown
- BioFLX Crown (Experimental): Experimental: BioFLX Crowns. In this split-mouth design, subjects were randomly assigned to receive BioFLX crowns on the side opposite of the 3M Stainless Steel Crowns.
  Interventions: Device: BioFLX crown

INTERVENTIONS:
Device: BioFLX crown — Device: BioFLX crown
  Arms: BioFLX Crown
Device: 3M Stainless Steel Crown — 3M Stainless Steel Crown
  Arms: SSC

SUMMARY:
The main reason for this research study is to learn more about a new flexible white dental crown (BioFLX) by comparing it to an existing flexible metal crown (Stainless Steel Crown). It is of interest to see if this new white crown is clinically equivalent to the existing silver crown that is mainly used in pediatric dentistry. A potential participant for this study would have cavities that require a crown, a type of filling that covers the entire tooth, and recommended dental work be done under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* CCHMC pediatric dental patients between the ages of 2 years to 5 years and 11 months, at the time of recruitment, who present to any CCHMC dental clinic location and then are found to need full mouth dental rehabilitation.
* Patients who speak the most common languages at CCHMC will be able to be recruited for the study.

  o English, Spanish, Arabic, Uzbek, Nepali, Chinese Mandarin, Russian, French.
* These patients must qualify for treatment at the CCHMC dental in-office general anesthesia (IOGA) area or the Procedure Center (PC). IOGA and the PC will be selected as a venue of treatment to control behavioral factors. This is not specific to the study and would occur due to their treatment needs.
* Participants will have at least one pair of contralateral primary molars with the need for a full coverage restoration in the same arch.

  * For example, tooth A & J, B & I, S & L, or T & K
  * For each participant, a minimum of one SSC or one PRC will be randomly assigned via a split mouth design to be placed as part of the study.
* Need for Full coverage and high caries risk will be defined by AAPD Best Practice Guidelines 2,16

  o Teeth With
  1. Extensive caries
  2. Cervical decalcification
  3. Developmental defects (e.g., hypoplasia, hypocalcification)
  4. When failure of other available restorative materials is likely (e.g., interproximal caries extending beyond line angles, patients with bruxism)
  5. Following pulpotomy or pulpectomy
  6. For definitive restorative treatment for high caries-risk children as defined by the AAPD
  7. For patients who exhibit high caries risk and whose treatment is performed under sedation or general anesthesia. This would be normal and not specific to the study.
* Participants who consent to the study, and who can be available for follow-up recall appointments.
* All participants will be ASA I or ASA II as defined by the American Society of Anesthesiologists.15

Exclusion Criteria:

* Participants who do not meet inclusion criteria will be excluded.

  * Participants whose teeth do not meet the inclusion criteria.
  * Participants who do not wish to participate in the study.
  * Patients who do not wish to or cannot reliably return for follow-up visits.
  * Red dye allergy as patient will not be able to be plaque disclosed during follow-up visits.
  * Participants who do not speak English, Spanish, Arabic, Uzbek, Nepali, Chinese Mandarin, Russian, French.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
The United States Public Health Service Restorative criteria | 36 months
  Study criteria being selected would be: Gingival Health, Plaque retention, Occlusal wear, and crown retention as defined by the following Alpha, Bravo, Charlie.
  Gingival Health according to the Modified Gingival Index (MGI):
  Alpha (A) normal gingiva
  Bravo (B) mild inflammation:
  Charlie (C) moderate inflammation
  Plaque Retention according to the Simplified Oral Hygiene Index (OHI -S):
  Alpha (A) 0, 1 Bravo (B)2 Charlie (C) 3
  Occlusal Wear:
  Alpha (A) occlusal surface intact Bravo (B) wear of occlusal surface without tooth surface exposure Charlie (C) wear of occlusal surface with tooth surface exposure.
  Crown retention:
  Alpha (A) Intact crown Bravo (B) partial loss of crown material Charlie (C) Crown lost

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
It can be if needed